## Appendix

Average how severe (0 –10)?

| Chronic Headache After Dural Puncture |
|---|
| Questionnaire (IRB 0335-18-SZMC) |
| Hello, my name is Dr |
| Informed Consent |
| We are conducting a research survey to better understand possible outcomes that women have after anesthesia for childbirth. We will be asking you a few questions about headache and backache based on your experience. With your permission, we will also look at your medical recordsfor things that might make it more or less likely that you would suffer from a headache or backache. We hope that your answers will help us to better treat other women with similar experiences. Your responses and identity will be kept confidential, your name and medical record number will be eliminated and only a number assigned to you. There are no risks to you, you may choose not to participate, your participation is voluntary, and refusal to participate will not affect your future care in any way. This will take approximately 5 to 10 minutes of your time. If you have any questions about the research, you may contact Prof. loscowich office at 02-6555104. |
| Yes: continue |
| No: Thank you very much for your time, have a great day! |
| 1. Did you have headaches or back pain before your delivery? |
| Yes: headache |
| On average how often did you have a headache? |
| Average how severe (0 –10)? |
| On average how long did they last? |
| How long have you had this problem? |
| Yes: backache |
| On average how often did you have back pain? |

On average how long did it last?

How long did you have this problem?

2. Have you had headaches since your delivery?

If Yes: headache questionnaire

3. Have you had back pain since your delivery?

If Yes: backache questionnaire

Last question

4. Can you give us a rating of your overall satisfaction

with your anesthesia care at Shaare Zedek Medical Center? (0 –10)

Thank you for helping us with this important research.

## Low Back Pain Rating Scale (Manniche et al.(5))

- 1. Pain at this time (0-10)
- 2. Worst back pain in 2 weeks (0 –10)
- 3. Average level of back pain (0 −10)

## **Disability Index**

- 1. Can you sleep at night without low back pain interfering?
- 2. Can you do your daily work without low back pain reducing your activities?
- 3. Can you do easy chores at home such as watering flowers or cleaning the table?
- 4. Can you put on shoes and stockings by yourself?
- 5. Can you carry 2 full shopping bags (10 kg in total)?
- 6. Can you get up from a low armchair without difficulty?

- 7. Can you bend over the wash basin to brush your teeth?
- 8. Can you climb stairs from one floor to another without resting because of low back pain?
- 9. Can you walk 400 meters without resting because of low back pain?
- 10. Can you run 100 meters without resting because of low back pain?
- 11. Can you ride a bike or drive a car without feeling any low back pain?
- 12. Does low back pain influence your emotional relationship to your nearest family?
- 13. Did you have to give up contact with other people within the last 2 weeks because of low back pain?
- 14. If it was of present interest, do you think that there are certain jobs which you would not be able to manage because of your back trouble?
- 15. Do you think that the low back pain will influence your future?

The Chronic Pain Grade Questionnaire (Smith et al.(6))

## For the following questions with a scale of 1-10 please circle one number only

| 10 is "pa | | | | | 1-10 sc | cale at t | he pres | ent tir | ne, that | is rig | tht now, where 0 is "no pain" and | l |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1015 P | No pain | | | | | | | | Pain as bad<br>as could be | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | 2. In the past six months, how intense was your worst pain rated on a 0-10 scale where 0 is "no pain" and 10 is "pain as bad as could be"? | | | | | | | | | | | |
| | No<br>pain | | | | | | | Pain as bad<br>as could be | | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| 3. In the past six months, on average, how intense was your pain rated on a 1-10 scale, where 0 is "no pain" and 10 is "pain as bad as could be"? (That is, your usual pain at times you were experiencing pain.) | | | | | | | | | | | | |
| | No<br>pain | | | | | | | | | | Pain as bad<br>as could be | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| 4. About how many days in the last six months have you been kept from your usual activities (work, school or housework) because of this pain? | | | | | | | | | | | | |
| | | | | | | | | | days | | | |
| | | | | | | | | | 7-14 days<br>15-30 days | | | |
| | | | | | | | | _ | | | | - |
| 5. In the past six months, how much has this pain interfered with your daily activities rated on a 1-10 scale where 0 is "no interference" and 10 is "unable to carry on activities"? | | | | | | | | | | | | |
| | | | | | | | | | your da | aily a | ctivities rated on a 1-10 scale who | ere |
| | interfer<br>No | | | | | | | | your da | aily a | ctivities rated on a 1-10 scale who<br>Unable to carry<br>on activities | ere |
| | interfer<br>No | ence" a | | | | | | | your da | aily a | Unable to carry | ere |
| 0 is "no | No<br>interfe<br>0 | ence" a<br>erence<br>1<br>x monti | nd 10 is<br>2<br>hs, how | "unabl | e to car | 5<br>pain ch | 6 anged | s"?<br>7<br>your a | 8<br>bility to | 9 | Unable to carry on activities | ere |
| 0 is "no | No<br>interfe<br>0 | ence" a<br>erence<br>1<br>x month | nd 10 is<br>2<br>hs, how | "unabl | e to car | 5<br>pain ch | 6 anged | s"?<br>7<br>your a | 8<br>bility to | 9 | Unable to carry<br>on activities | ere |
| 0 is "no | No interfer O e past si ctivities | ence" a<br>erence<br>1<br>x month | nd 10 is<br>2<br>hs, how | 3<br>much to change | e to car | 5<br>pain ch | 6<br>sanged y | s"?<br>7<br>your a | 8<br>bility to<br>e"? | 9 | Unable to carry on activities 10 part in recreational, social and Extreme | ere |
| 0 is "no 6. In the family a | No interfer O e past si ctivities No chang O e past si | erence 1 x monti s where 1 x monti | 2 hs, how 0 is "no | 3 much to change | 4 nas this 4 nas this | 5<br>pain ch<br>10 is "es | 6 sanged streme | 7<br>your a<br>chang | 8<br>bility to<br>e"? | 9<br>take | Unable to carry on activities 10 part in recreational, social and Extreme change | |
| 6. In the family a | No interfer O e past si ctivities No chang O e past si | erence 1 x month where te 1 x month to the | 2 hs, how 0 is "no | 3 much to change | 4 nas this 4 nas this | 5<br>pain ch<br>10 is "es | 6 sanged streme | 7<br>your a<br>chang | 8<br>bility to<br>e"? | 9<br>take | Unable to carry on activities 10 part in recreational, social and Extreme change | |